CLINICAL TRIAL: NCT03741933
Title: An Open-label, Single-Arm Pilot Study Investigating the Efficacy and Safety of Apremilast for the Treatment of Moderate to Severe Chronic Hand Dermatitis
Brief Title: Apremilast and Moderate to Severe Chronic Hand Dermatitis
Acronym: CHD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The principal investigator left George Washington University and closed the study at their departure.
Sponsor: George Washington University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP-CL-DERMAT-PI-13069
Record Dates: First submitted 2018-08-22; First posted 2018-11-15 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Chronic Hand Dermatitis
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Intervention Model Description: All participants will be patients that have been screened within the Department of Dermatology at the GW MFA. Individuals meeting inclusion and exclusion criteria will be enrolled into the study. A total of 10 patients will be enrolled in the study and each patient will be given Apremilast 30 mg twice daily to be administered for a period of 6 months. Patients will present to clinic for clinical assessments, adverse event monitoring, laboratory testing, and/or photography at the following time periods of therapy: baseline and 2 weeks, 4 weeks, and every 4 weeks thereafter until completion of the 6 month treatment period. Additionally, all patients will be required to return for a 4-week follow up visit after completing the final dose of the study medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apremilast (Experimental): 30 mg twice daily to be administered for a period of 6 months
  Interventions: Drug: Apremilast 30mg

INTERVENTIONS:
Drug: Apremilast 30mg — Apremilast 30 mg tablet
  Other Names: Otezla; CC-10004

SUMMARY:
Investigators have designed a pilot study involving chronic hand dermatitis (CHD) patients who attend the dermatology clinic at the George Washington Medical Faculty Associates (GW MFA) in order to assess the efficacy and safety of apremilast treatment for the treatment of moderate to severe CHD.

DETAILED DESCRIPTION:
Hand dermatitis is one of the most common skin disorders encountered by dermatologists. Chronic hand dermatitis (CHD) is often due to allergic contact dermatitis (ACD) or irritant contact dermatitis (ICD) and has a 1-year and lifetime prevalence of up to 10% and 15%, respectively, in the general population. On average, the disease affects patients for about 7 to 11 years.

Patients with ACD show an increase in cytokines produced from T helper (Th)1 and Th17 cells, including (interleukin) IL-17 and IL-23, which are also implicated in the pathogenesis of psoriasis. Apremilast, a small molecule phosphodiesterase-4 (PDE-4) inhibitor, has demonstrated clinical efficacy and tolerability in the treatment of psoriasis and psoriatic arthritis, likely through the blockade of IL-17, IL-23, and several other pro-inflammatory mediators. Therefore, it may provide an effective treatment option for other Th1 and Th17-mediated disease (such as CHD due to ACD and ICD), which share a common immunologic pathway with psoriasis. Investigators hypothesize that apremilast has the ability to decrease disease severity in patients with moderate-to-severe CHD that is either secondary to psoriasis, or occurring in patients with an atopic or allergic past medical history. Hence, investigators have designed a pilot study involving CHD patients who attend the dermatology clinic at the George Washington Medical Faculty Associates (GW MFA) in order to assess the efficacy and safety of apremilast treatment for the treatment of moderate to severe CHD. The objectives are as follows:

Primary objective:

1. To evaluate the efficacy of Apremilast 30mg twice daily administered as monotherapy in the treatment of moderate-to-severe CHD as assessed by improvement of the Physician Global Assessment (PGA).

Secondary objectives:

1. To evaluate the safety and tolerability of Apremilast 30mg twice daily as assessed by monitoring adverse events, laboratory values (CBC, CMP), and physical examination.
2. To evaluate CHD lesion time to response (TTR) as assessed by Modified Total Lesion Symptom Score (mTLSS).
3. To evaluate the patient's perception of CHD severity improvement as assessed by the Patient Global Assessment (PaGA).
4. To evaluate the patient's health-related quality of life as assessed by the Dermatology Life Quality Index (DLQI) questionnaire a measurement of the patient's subjective symptoms.

STUDY ENDPOINTS

Primary endpoint:

1. Proportion of patients achieving a 2 point decrease in Physician Global Assessment (PGA) at the end of the study.

Secondary endpoints:

1. Proportion of patients achieving Physician Global Assessment (PGA) score of 0 (clear) or 1 (almost clear) at end of study.
2. Change in mTLSS, patient global assessment, and DLQI scores from baseline to end of study.
3. Photographic improvement of CHD from baseline to end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 18-79 years.
2. Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
3. Clinical diagnosis of CHD as defined by hand dermatitis for more than 6 months or more than 2 flares within 12 months.
4. Moderate to severe CHD, defined as a PGA score of 3 (moderate) or 4 (severe).
5. History of AD, childhood eczema, ACD, or ICD.
6. History of disease that is unresponsive to conventional treatment (i.e. corticosteroids, calcineurin inhibitors, phototherapy) for CHD. Lack of response to treatment is defined as an unsatisfactory outcome (no response, transient response to ongoing treatment or lack of tolerability) based on patient history and medical records.
7. No other active skin diseases or acute skin infections dominating the clinical picture.
8. Females of childbearing potential (FCBP)† must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive§ options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy;

OR

Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

† A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been postmenopausal for at least 24 consecutive months (that is, has had menses at any time during the preceding 24 consecutive months).

§ The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).

Exclusion Criteria:

1. <18 or >79 years of age.
2. Evidence of tinea mannum involving the hands (verified by positive fungal culture).
3. Evidence of an active untreated infection (bacterial, fungal, viral etc) involving the hands at baseline visit.
4. Use of topical corticosteroids on the hands within 2 weeks prior to baseline visit.
5. Use of topical calcineurin inhibitor (tacrolimus, pimecrolimus) on the hands within 2 weeks prior to baseline visit.
6. Use of crisaborole on the hands within 2 weeks prior to baseline visit.
7. Use of light based treatments on the hands within 1 month prior to baseline visit.
8. Use of systemic therapy (cyclosporine, azathioprine, methotrexate, alitretinoin) within 4 weeks prior to the start of study medication OR 5 pharmacokinetic / pharmacodynamics half-lives (whichever is longer).
9. Inability to make study visits or anticipated poor compliance.
10. Pregnant females or nursing mothers. Eligible women of reproductive age will be required to adhere to strict pregnancy prevention measures, which includes a negative urine pregnancy test at screening and subsequent visits.
11. History of Tuberculosis, Hepatitis B, C, or HIV.
12. Any history or evidence of a medical comorbidity that would make the subject, in the opinion of the investigator, unsuitable for the study.
13. Active substance abuse or a history of substance abuse within 6 months prior to Screening.
14. Other than disease under study, any clinically significant (as determined by the Investigator) cardiac, endocrinology, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled.
15. Life threatening illness that would interfere with the subject's ability to complete the study.
16. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study.
17. Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years.
18. Malignancy or history of malignancy, except for:

    1. Treated [i.e., cured] basal cell or squamous cell carcinomas of the skin with no evidence of recurrence within the previous 5 years.
    2. Treated [i.e., cured] cervical intraepithelial neoplasia (CIN) or carcinoma in situ of cervix with no evidence of recurrence within the previous 5 years.
19. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer).
20. Prior treatment with apremilast.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of Apremilast 30mg twice daily administered as monotherapy in the treatment of moderate-to-severe CHD as assessed by improvement of the Physician Global Assessment (PGA). | 24 weeks
  PGA classifies the severity of CHD into five categories (clear, almost clear, mild, moderate, and severe). The PGA scale ranges from 0 (no symptoms) to 4 (severe disease). PGA ratings will be based on an integrated clinical picture of signs, symptoms, and the extent of disease.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of Apremilast 30mg twice daily through incidence of adverse events. | 24 weeks
  Evaluation of all adverse events from Day 0 to Week 24.
To evaluate CHD lesion time to response (TTR) as assessed by Modified Total Lesion Symptom Score (mTLSS). | 24 weeks
  The mTLSS is a 4-point scale that is calculated as sum of assigned scores for the symptoms of erythema, scaling, lichenification/hyperkeratosis, vesiculation, edema, fissures and pruritus/pain. The total score ranges from 0 (best) to 21 (worst). Scores will be assigned for the most affected side (palmar or dorsal) of the most affected hand. The investigator will assign mTLSS scores for patients at all visits.
To evaluate the patient's perception of CHD severity improvement as assessed by the Patient Global Assessment (PaGA). | 24 weeks
  Patients will be asked by the investigator to grade their overall change from baseline by selecting one of the following descriptions, which best matches their perception of overall treatment effect: cleared or almost clear (at least 90% clearing), marked improvement (at least 75% clearing), moderate improvement (at least 50% clearing), mild improvement (at least 25% clearing), no change, or worsening.
To evaluate the patient's health-related quality of life as assessed by the Dermatology Life Quality Index (DLQI) questionnaire a measurement of the patient's subjective symptoms. | 24 weeks
  The DLQI is a 10-item, validated questionnaire used to assess the impact of dermatitis disease symptoms and treatment on quality of life (QOL). Patients are asked to assess QOL over the past week with a simple response (0 to 3; where 0 = "not at all" and 3 = "very much"), with an overall scoring system of 0 to 30 and a high score being indicative of a poor QOL.

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Department of Dermatology, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Coenraads PJ. Hand eczema. N Engl J Med. 2012 Nov 8;367(19):1829-37. doi: 10.1056/NEJMcp1104084. PMID 23134383
- [Background] Menne T, Johansen JD, Sommerlund M, Veien NK; Danish Contact Dermatitis Group. Hand eczema guidelines based on the Danish guidelines for the diagnosis and treatment of hand eczema. Contact Dermatitis. 2011 Jul;65(1):3-12. doi: 10.1111/j.1600-0536.2011.01915.x. PMID 21658053
- [Background] English J, Aldridge R, Gawkrodger DJ, Kownacki S, Statham B, White JM, Williams J. Consensus statement on the management of chronic hand eczema. Clin Exp Dermatol. 2009 Oct;34(7):761-9. doi: 10.1111/j.1365-2230.2009.03649.x. PMID 19747339
- [Background] Berg S. Prävalenz von Handekzemen in Heidelberg und weltweit - die Heidelberger Prävalenzstudie im Vergleich mit Ergebnissen aus der Literatur. Dissertation, Heidelberg, 2005
- [Background] Hald M, Berg ND, Elberling J, Johansen JD. Medical consultations in relation to severity of hand eczema in the general population. Br J Dermatol. 2008 Apr;158(4):773-7. doi: 10.1111/j.1365-2133.2007.08431.x. Epub 2008 Jan 30. PMID 18241259
- [Background] Brunner PM, Leung DYM, Guttman-Yassky E. Immunologic, microbial, and epithelial interactions in atopic dermatitis. Ann Allergy Asthma Immunol. 2018 Jan;120(1):34-41. doi: 10.1016/j.anai.2017.09.055. Epub 2017 Nov 7. PMID 29126710
- [Background] Bissonnette R, Haydey R, Rosoph LA, Lynde CW, Bukhalo M, Fowler JF, Delorme I, Gagne-Henley A, Gooderham M, Poulin Y, Barber K, Jenkin P, Landells I, Pariser DM. Apremilast for the treatment of moderate-to-severe palmoplantar psoriasis: results from a double-blind, placebo-controlled, randomized study. J Eur Acad Dermatol Venereol. 2018 Mar;32(3):403-410. doi: 10.1111/jdv.14647. Epub 2017 Nov 15. PMID 29055155